CLINICAL TRIAL: NCT01086072
Title: Survival Trends in Myocardial Infarction 1994 - 2010
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Sponsor
Other Study IDs: ELD003
Record Dates: First submitted 2010-03-08; First posted 2010-03-12 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2010-03

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Myocardial Infarction - STEMI
- Myocardial Infarction - NSTEMI

SUMMARY:
Practice in management of myocardial ischemia and infarction has changed significantly over the past 20 years, both in terms of immediate management and secondary prevention.

The aim of this observational study is to utilize the established record linkage data available in Tayside to investigate the trends in survivors of myocardial infarction in Tayside since 1994.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial Infarction

Exclusion Criteria:

* Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with Myocardial Infarction in Tayside 1994 - 2010
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2010-03-01 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2011-03-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Mortality | 20 years
  All cardiovascular mortality

SECONDARY OUTCOMES:
Cardiovascular hospitalisation | 20 years
  Hospitalisation for cardiovascular cause after initial presentation

CONTACTS AND LOCATIONS:
Locations (1):
- Douglas Elder, Dundee, United Kingdom